CLINICAL TRIAL: NCT01055652
Title: An Open-label, Multi-centre, Drug-drug Interaction Study to Assess the Effect of Voglibose (0.2 mg Tid) on the Pharmacokinetics, Safety and Tolerability of Single Oral Administration of Dapagliflozin (10 mg) in Japanese Patients With Type 2 Diabetes
Brief Title: Drug-drug Interaction Study of Dapagliflozin With Voglibose in Japanese Type 2 Diabetes Mellitus Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: D1692C00002
Record Dates: First submitted 2010-01-22; First posted 2010-01-25 (Estimated); Last update posted 2011-10-17 (Estimated); Status verified 2010-10

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes mellitus; Japanese; phase 1; safety; dapagliflozin; Pharmacokinetics; Drug-drug Interaction; voglibose
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Dapagliflozin

INTERVENTIONS:
Drug: Dapagliflozin — 10mg, oral, once daily

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics of dapagliflozin when administered alone or in combination with voglibose in Japanese patients with type 2 diabetes by assessment of AUC and Cmax of dapagliflozin

ELIGIBILITY:
Inclusion Criteria:

* Already on voglibose treatment with a steady dosage for at least 8 weeks
* Provision of informed consent prior to any study specific procedures
* Diagnosed with type 2 diabetes

Exclusion Criteria:

* Having clinically relevant medical history or concurrent disease such as cardiovascular disease, renal disease, retinopathy, hepatic disease and haematological disease.
* The investigator(s)judged that the Subject should not participate in the study according to screening test or medical history.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-01; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
To evaluate the pharmacokinetics of dapagliflozin when administered alone or in combination with voglibose in Japanese patients with type 2 diabetes by assessment of AUC and Cmax of dapagliflozin | Plasma samples will be collected through Visit 4 (up to 72 hours = 3 days after dose) for PK assessment for period 1. Plasma samples will be collected through Visit 7 (up to 72 hours = 3 days after dose) for PK assessment for period 2.

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of dapagliflozin when administered alone or in combi-nation with voglibose in Japanese patients with type 2 diabetes. | Plasma samples will be collected through Visit 4 (up to 72 hours = 3 days after dose) for PK assessment for period 1. Plasma samples will be collected through Visit 7 (up to 72 hours = 3 days after dose) for PK assessment for period 2.
To evaluate the pharmacokinetics of dapagliflozin when administered alone or in combination with voglibose in Japanese patients with type 2 diabetes by assessmentof AUC0-t, tmax, t1/2, CL/F. | Plasma samples will be collected through Visit 4 (up to 72 hours = 3 days after dose) for PK assessment for period 1. Plasma samples will be collected through Visit 7 (up to 72 hours = 3 days after dose) for PK assessment for period 2.

CONTACTS AND LOCATIONS:
Overall Officials: Nobuyuki Shiga, Study Director — AstraZeneca
Locations (2):
- Japan (2):
  - Research Site, Moriya
  - Research Site, Osaka